CLINICAL TRIAL: NCT04727112
Title: Asthma and Allergy Screening AA2000 (Cross Sectional)
Acronym: AA2000
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Vibeke Backer, Professor, Bispebjerg Hospital
Other Study IDs: asthma and allergy screening
Record Dates: First submitted 2013-11-05; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Asthma
Keywords: asthma; airway hyperresponsiveness; asthma management
MeSH Terms: conditions — Asthma; Respiratory Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- asthma and rhinitis: Screening of patients with upper and lower airway symptoms
  Interventions: Drug: Usual care versus primary care
- asthma and rhintis follow-up: same Group as screened in 2000, was followed up three years later
  Interventions: Drug: Usual care versus primary care

INTERVENTIONS:
Drug: Usual care versus primary care — RCT study
  Other Names: RCT study, usuar care in specialist setting (GINA and ARIA)

SUMMARY:
Asthma screening of 493 asthma patients

DETAILED DESCRIPTION:
Questionnaire, and testing

ELIGIBILITY:
Inclusion Criteria: respiratory symptoms suggestive for asthma -

Exclusion Criteria:COPD

-

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Population based asthma study
Sampling Method: Probability Sample
Enrollment: 493 (Actual)
Dates: Start 2000-01; Primary Completion 2003-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
ACQ | 2004
  Questionnaire based
AQLQ | 2004
  Questionnaire based

SECONDARY OUTCOMES:
FEV1 | 2004
  Lung function

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Backer, MD, Principal Investigator — Bispebjerg Hospital